CLINICAL TRIAL: NCT04277637
Title: A Phase 1a/1b Open-Label Dose Escalation and Expansion Study of Bcl-2 Inhibitor BGB-11417 in Patients With Mature B-Cell Malignancies
Brief Title: Study of Bcl-2 Inhibitor Sonrotoclax (BGB-11417) in Participants With Mature B-Cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-101; 2024-515592-35-00 (EU CTIS Number); 2020-004641-37 (EudraCT Number)
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Mature B-Cell Malignancies
Keywords: NHL; BCL2 Inhibitor; CLL; MCL; MZL; SLL; WM; Bcl-2i; BTKi
MeSH Terms: interventions — zanubrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sonrotoclax Monotherapy Dose Finding: Part 1 (Experimental): Participants with relapsed/refractory (R/R) non-Hodgkin lymphoma (NHL) including follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), marginal zone lymphoma (MZL) or transformed NHL, mantle cell lymphoma (MCL); Waldenströms macroglobulinemia (WM); and chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) will receive oral sonrotoclax evaluated as monotherapy.
  Interventions: Drug: Sonrotoclax
- Sonrotoclax Monotherapy Expansion Cohorts: Part 2 (Experimental): Participants with R/R indolent NHL including FL, MZL; aggressive NHL including DLBCL, transformed NHL; CLL/SLL with low tumor burden or low creatine clearance; CLL/SLL with without high tumor burden or low creatine clearance will receive oral sonrotoclax at the RP2D dose to further define the safety profile.
  Interventions: Drug: Sonrotoclax
- Sonrotoclax + Zanubrutinib Combination Therapy Dose Finding: Part 3 (Experimental): Participants with R/R MCL, R/R or treatment-naïve (TN) CLL/SLL will receive oral sonrotoclax in combination with zanubrutinib.
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib
- Sonrotoclax + Zanubrutinib Combination Therapy Dose Expansion: Part 4 (Experimental): Participants with R/R indolent NHL including FL, MZL; aggressive NHL including DLBCL, transformed NHL; R/R MCL; R/R or treatment-naïve (TN) CLL/SLL will receive oral sonrotoclax in combination with zanubrutinib at an RP2D dose to further define the safety profile.
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib
- Sonrotoclax + Zanubrutinib Combination Therapy Dose Escalation: Part 5 (Experimental): Participants with treatment naïve CLL/SLL will receive oral sonrotoclax in combination with obinutuzumab without and with zanubrutinib.
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib; Drug: Obinutuzumab
- Sonrotoclax + Zanubrutinib Combination Therapy Dose Expansion: Part 6 (Experimental): Participants with treatment naïve CLL/SLL will receive oral sonrotoclax in combination with obinutuzumab without and with zanubrutinib at an RP2D dose to further define the safety profile.
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Sonrotoclax — Film-coated tablets administered once daily at a dose as specified in the treatment arm
  Other Names: BGB-11417
Drug: Zanubrutinib — 320 mg daily administered as two 80-mg capsules twice a day (160 mg twice a day) or as four 80-mg capsules once a day (320 mg once a day)
  Other Names: BGB-3111
  Arms: Sonrotoclax + Zanubrutinib Combination Therapy Dose Escalation: Part 5; Sonrotoclax + Zanubrutinib Combination Therapy Dose Expansion: Part 4; Sonrotoclax + Zanubrutinib Combination Therapy Dose Expansion: Part 6; Sonrotoclax + Zanubrutinib Combination Therapy Dose Finding: Part 3
Drug: Obinutuzumab — Given as an intravenous infusion administered per label.
  Arms: Sonrotoclax + Zanubrutinib Combination Therapy Dose Escalation: Part 5; Sonrotoclax + Zanubrutinib Combination Therapy Dose Expansion: Part 6

SUMMARY:
The purpose of this study is to determine the safety, tolerability; and to define the maximum tolerated dose (MTD) and Recommended Phase 2 Dose (RP2D); and to evaluate the safety and tolerability of the ramp-up dosing schedule and at the RP2D of BGB-11417 monotherapy, and when given in combination with zanubrutinib and obinutuzumab.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of one of the following:

NHL Cohorts:

1. MZL i. R/R extranodal, splenic, or nodal MZL defined as disease that relapsed after, or was refractory to, at least one prior therapy ii. Active disease requiring treatment
2. FL i. R/R FL (Grade 1, 2 or 3a based on the WHO 2008 classification of tumors of hematopoietic and lymphoid tissue) and defined as disease that relapsed after, or was refractory to, at least 1 prior systemic therapy
3. DLBCL i. R/R DLBCL (including all subtypes of DLBCL) defined as disease that relapsed after, or was refractory to, at least two prior systemic therapies and has either progressed following or is not a candidate for autologous stem cell transplant (due to comorbidities or non-responsiveness to salvage chemotherapy)
4. Transformed indolent B-cell NHL i. Any lymphoma otherwise eligible for Part 1 that has transformed into a more aggressive lymphoma. Patients with transformation from CLL or SLL (Richter's transformation) are not eligible for Part 1

   CLL/SLL Cohorts:
5. CLL/SLL diagnosis that meets the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria i. Disease characterized as Treatment Naive (TN) or R/R disease defined as disease that relapsed after, or was refractory to, at least 1 prior therapy ii. Requiring treatment as defined by history

   MCL cohorts:
6. WHO-defined MCL i. R/R MCL defined as disease that relapsed after, or was refractory to, at least 1 prior systemic therapy; ii. Requiring treatment in the opinion of the investigator

WM cohorts:

g. WHO-defined WM (clinical and definitive histologic diagnosis) i. R/R disease defined as disease that relapsed after, or was refractory to, at least 1 prior therapy; ii. Meeting at least 1 criterion for treatment according to consensus panel criteria from the Seventh International Workshop on Waldenström's Macroglobulinemia (Dimopoulos et al 2014)

* Measurable disease by computed tomography (CT)/magnetic resonance imaging (MRI), defined as:

  1. CLL: at least 1 lymph node > 1.5 cm in longest diameter and measurable in 2 perpendicular dimensions or clonal lymphocytes measured by flow cytometry
  2. DLBCL, FL, MZL, MCL, or SLL: at least 1 lymph node > 1.5 cm in longest diameter OR 1 extranodal lesion > 1.0 cm in the longest diameter, measurable in at least 2 perpendicular dimensions. For MZL, isolated splenomegaly is considered measurable for this study
  3. WM: serum immunoglobulin (Ig) M level > 0.5 g/dL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Adequate organ function
* Adequate pancreatic function indicated by:

  1. Serum amylase ≤ 1.5 x upper limit of normal (ULN)
  2. Serum lipase ≤ 1.5 x ULN

Key Exclusion Criteria:

* Known current central nervous system involvement by lymphoma/leukemia
* Known plasma cell neoplasm, prolymphocytic leukemia, history of or currently suspected Richter's syndrome
* Prior therapy ≥ 2 months with or progression on a B-cell lymphoma-2 (Bcl-2) inhibitor

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment Emergent Adverse Events (TEAEs) | Up to 30 days after the last dose of study drug, an average of 18 months
Number of Participants Experiencing Serious Adverse Events (SAEs) | Up to 30 days after the last dose of study drug, an average of 18 months
Number of Participants Experiencing Adverse Events (AEs) leading to discontinuation of Sonrotoclax | Up to 30 days after the last dose of study drug, an average of 18 months
Part 1, Part 3: Maximum Tolerated Dose (MTD) of Sonrotoclax | Up to approximately 2 months
Part 1, Part 3, Part 5: RP2D of Sonrotoclax | Day 1 to last dose of study drug, an average of 18 months
Part 1, Part 3, Part 5: Number of participants experiencing tumor lysis syndrome (TLS) relevant events | Up to 30 days after the last dose of study drug, an average of 18 months
Part 1, Part 3, Part 5: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs | Up to approximately 2 months

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) After a Single Dose of Sonrotoclax | Predose up to 12 hours postdose
Area Under the Concentration-Time Curve from Time 0 to the Last Quantifiable Concentration (AUC0-last) After a Single Dose of Sonrotoclax | Predose up to 12 hours postdose
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-∞) After a Single Dose of Sonrotoclax | Predose up to 12 hours postdose
Time Taken for Half the Initial Dose Administered to Be Eliminated from The Body (T1/2) of Sonrotoclax | Predose up to 12 hours postdose
Time to Maximum Plasma Concentration (Tmax) After a Single Dose of Sonrotoclax | Predose up to 12 hours postdose
Apparent Clearance (CL/F) After a Single Dose of Sonrotoclax | Predose up to 12 hours postdose
Apparent volume of distribution (Vz/F) After a Single Dose of Sonrotoclax | Predose up to 12 hours postdose
Steady State Area Under the Concentration-Time Curve of 0 - Last Day (AUCLast, ss) of Sonrotoclax | Predose up to 12 hours postdose
Part 3, Part 4: Steady State Area Under the Concentration-Time Curve of 0 - Last Day (AUCLast, ss) of zanubrutinib | Predose up to 12 hours postdose
Steady State Maximum Observed Plasma Concentration (Cmax, ss) of Sonrotoclax | Predose up to 12 hours postdose
Part 3, Part 4: Steady State Maximum Observed Plasma Concentration (Cmax, ss) of zanubrutinib | Predose up to 12 hours postdose
Steady State Trough Observed Plasma Concentration (Ctrough, ss) of Sonrotoclax | Predose up to 12 hours postdose
Part 3, Part 4: Steady State Trough Observed Plasma Concentration (Ctrough, ss) of zanubrutinib | Predose up to 12 hours postdose
Steady State Time to Maximum Plasma Concentration (Tmax, ss) of Sonrotoclax | Predose up to 12 hours postdose
Part 3, Part 4: Steady State Time to Maximum Plasma Concentration (Tmax, ss) of zanubrutinib | Predose up to 12 hours postdose
Part 2: AUC of Sonrotoclax administered after a high fat/calorie meal (HF-Fed) | Predose up to 12 hours postdose
Part 2: Cmax of Sonrotoclax administered after a high fat/calorie meal (HF-Fed) | Predose up to 12 hours postdose
Part 2, Part 4, Part 6: Overall Response Rate (ORR) as Assessed by the Investigator | Up to 18 months
  ORR is defined as the proportion of participants who had confirmed complete response Complete Response (CR) or Partial Response (PR)
Part 2: Major Response Rate (MRR) for WM as Assessed by the Investigator | Up to 18 months
Part 6: Minimum residual disease (MRD) negativity as measured by next generation sequencing | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (44):
- United States (13):
  - UCLA Hematologyoncology, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - John Theurer Cancer Center Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - The James Cancer Hospital and Solove Research Institute At Ohio State University, Columbus, Ohio
  - Upmc Hillman Cancer Center(Univ of Pittsburgh), Pittsburgh, Pennsylvania
  - Md Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (12):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Orange Health Service (Central West Cancer Care Centre), Orange, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - John Flynn Private Hospital, Tugun, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford PK, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Universitatsklinikum Carl Gustav Carus An Der Technischen Universitat Dresden, Dresden, Germany
- Italy (6):
  - Ospedale San Raffaele, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale Santa Maria Della Misericordia, Perugia
  - Azienda Unita Sanitaria Locale Di Ravenna, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Centroricerche Cliniche Di Verona Srl, Verona
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - North Shore Hospital, Takapuna
  - Wellington Regional Hospital (Ccdhb), Wellington
- Spain (8):
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Vall D Hebron Institute of Oncology Vhio, Barcelona
  - Ico H Duran I Reynals, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Start Madrid Fundacion Jimenez Diaz, Madrid
  - Clinica Universidad de Navarra Pamplona, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
- The Leeds Teaching Hospitals Nhs Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/